CLINICAL TRIAL: NCT04284488
Title: A Phase Ib/II Clinical Study to Evaluate the Efficacy and Safety of APG-1387 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: Dose-escalation Study of APG-1387 and Toripalimab in Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Strategy
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG1387XC101
Record Dates: First submitted 2020-02-05; First posted 2020-02-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — APG-1387; Injections; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APG-1387 in combination with Toripalimab (Experimental)
  Interventions: Drug: APG-1387 for Injection; Drug: Toripalimab

INTERVENTIONS:
Drug: APG-1387 for Injection — APG-1387 IV on Days 1 and 8 of each 21-Day Cycle. The following doses of APG-1387 to be studied: 20, 30, and 45mg. In the phase II, the assigned recommended phase two dose will be administered in all cohorts.
Drug: Toripalimab — 240 mg toripalimab IV on Day 1 of each 21-Day Cycle
  Other Names: JS001

SUMMARY:
An ascending dose study in patients with solid tumors to evaluate the safety, tolerability, pharmacodynamics and efficacy of APG-1387 in combination with toripalimab. A phase II study of 3 cohorts will be included.

DETAILED DESCRIPTION:
This study will be conducted in two phases. In phase Ib, the safety and efficacy of different dose levels of APG-1387 in combination with 240 mg toripalimab will be explored to determine the recommended Phase 2 dose (RP2D) of APG-1387 in combination therapy, both administered as a 30-minute intravenous (IV) infusion. The following proposed doses of APG-1387 are to be evaluated: 20,30, or 45mg .

The Phase II portion, will compromise 3 cohorts of 15-25 patients.

The 3 cohorts will include the following:

* Colorectal cancer
* Nasopharyngeal carcinoma
* Non-small cell lung cancer with PD-1 antibody refractory or relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed advanced solid tumors

   1. For phase II CRC group only: Patients with histologically confirmed microsatellite stable (detected by immunohistochemistry, PCR or NGS methods) advanced colorectal cancer.
   2. For phase II NPC group only: Patients with histologically or cytologically confirmed advanced NPC.
   3. For phase II NSCLC group only: Patients with histologically confirmed or cytologically confirmed advanced non-small cell lung cancer together with wild-type EGFR/ALK/ROS1 (first or second-generation sequencing results are allowed).
2. Patients who have failed standard antitumor therapy.
3. At least one evaluable lesion according to RECIST 1.1 criteria.
4. Age greater than 18 years, both men and women.
5. ECOG: 0 to 1.
6. Expected survival ≥ 3 months.
7. The function of vital organs meets the following criteria (no blood components and cell growth factors are allowed 2 weeks before the start of study treatment):

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   2. Platelets ≥ 100 × 10^9/L;
   3. Hemoglobin ≥ 90 g/L;
   4. Serum albumin ≥ 30 g/L;
   5. Total bilirubin ≤ 1.5 x the upper limit of normal(ULN), ALT and AST ≤ 2.5 x ULN; if there is liver metastasis, ALT and AST ≤ 5 x ULN;
   6. Serum creatinine ≤ 1.5 x ULN ; or if Serum creatinine >1.5 x UL, 24-hour creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula);
8. Patients with asymptomatic brain metastases (not requiring pharmacological control) or brain metastases that have been stable for more than 28 days after treatment.
9. Patients must have recovered to Grade 1 or less from adverse reactions resulting from prior antineoplastic therapy (except alopecia and sensory neuropathy not exceeding Grade 2).
10. Males, women of childbearing potential (postmenopausal women who must have been postmenopausal for at least 12 months to be considered of non-childbearing potential) and their partners voluntarily use contraception deemed effective by the investigator during treatment and for at least three months after the last dose of study drug.
11. Able to understand and voluntarily sign a written informed consent form, which must be signed prior to the performance of any trial-specified study procedures.
12. Patients must be voluntary and able to complete study procedures and follow-up examinations.

Exclusion Criteria:

1. Cytotoxic chemotherapy, radiation therapy, surgery (except minor surgery), anticancer therapy with hormone therapy (except hormone for hypothyroidism or estrogen replacement therapy (ERT)), or any clinical study treatment within 28 days prior to the first dose of study drug; or clinically significant tumor embolism or tumor lysis syndrome (TLS).
2. Immunotherapy, biologic therapy or anti-TNFa therapy within 28 days or 5 half-lives (whichever is shorter) prior to receiving the first dose of study drug.
3. Patients who have received targeted therapy within 28 days prior to first dose of study drug.
4. Prior treatment with anti PD-1, anti PD-L1, or anti PD-L2 agents (Phase II CRC cohort only).
5. Patients have an immunodeficiency diagnosis or are receiving chronic systemic steroid therapy (daily dose of more than 10 mg prednisone equivalent) or any form of immunosuppressive therapy 7 days prior to the first dose of trial treatment.
6. Patients have any active autoimmune disease or a history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, decreased thyroid function (can be included if hormone replacement therapy is effective); patients with vitiligo or asthma that has been completely relieved in childhood and does not require any intervention after adulthood can be included, and patients with asthma requiring bronchodilators for medical intervention cannot be included.
7. Patient has an active infection or unexplained fever > 38.5。C within 2 weeks prior to the first dose (subjects may be enrolled due to tumor generated fever as judged by the investigator).
8. Any evidence of a past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroids, or clinically active interstitial lung disease.
9. Hepatic decompensation.
10. Evidence of any severe or uncontrolled systemic disease; various chronic active infections such as hepatitis B (evidence of hepatitis activity such as HBV-DNA ≥ 104 copies/mL or 2000 IU/mL), hepatitis C, and HIV.
11. Any of the following cardiac criteria: Mean QTc> 470 msec at rest during screening; Any clinically important abnormality in rhythm, conduction, or morphology of the resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block); Congenital long QT syndrome or family history of long QT syndrome.
12. Uncontrolled hypertension (requiring 2 or more medications to control blood pressure); Unstable cardiac pain; Angina pectoris within 3 months of study entry; Congestive heart failure (NYHA class II or higher); Previous myocardial infarction (NSTEMI or STEMI) within 6 months of study entry; Serious cardiac arrhythmia requiring medical attention; Serious hepatic, renal, gastrointestinal, or metabolic disease.
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to APG-1387 or toripalimab or their constituents.
14. Have received a live vaccine within 28 days prior to the first dose of investigational product. Live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacille Calmette-Guérin vaccine (BCG) and typhoid. Injectable seasonal influenza vaccines are usually inactivated viral vaccines and are therefore allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed.
15. Patients who have not sufficiently recovered after surgical treatment as judged by the investigator. Patients with major surgery within 28 days prior to the first dose of study drug and minor surgery within 7 days prior to the start of the study.
16. Pregnant or lactating female patients.
17. The subject has other factors that may cause the subject to be forced to terminate the study, such as suffering from other serious diseases (including mental illness) requiring concomitant treatment, severe abnormalities in laboratory tests, family or social factors, conditions that may affect the safety of the subject or the collection of trial data, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 dose(RP2D) (Applicable for: phase I stage in various solid tumor types). | 21 days.
  Recommended phase 2 dose(RP2D) of APG-1387 in combination with toripalimab in subjects with solid tumors.
Disease control rate (Applicable for: phase II in cohorts of Colorectal Cancer, Nasopharyngeal Carcinoma and Non-Small Cell Lung Cancer) . | 18-24months.
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Version1.1 and iRECIST.

SECONDARY OUTCOMES:
Overall Response (Applicable for: phase I stage in various solid tumor types) | 18-24months.
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and iRECIST.
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) (Applicable for: phase II) | 18-24months.
  Patients treatment related adverse events (AEs) and severe adverse events (SAEs) will be assessed according NCI CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, M.D., Ph.D., Study Director — Ascentage Pharma Group Inc.
Locations (3):
- China (3):
  - Foshan First People's Hospital, Foshan, Guangdong
  - Sun-Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Hospital OF Guangxi Medical University, Nanning, Guangxi